CLINICAL TRIAL: NCT06423755
Title: Swimming Versus Standard Physiotherapy Care as Rehabilitation Modalities for Persistent Low Back Pain: A Feasibility Study
Brief Title: Swimming Versus Standard Physiotherapy Care as Rehabilitation Modalities for Persistent Low Back Pain: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 264307
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low-back Pain
Keywords: Rehabilitation; Swimming; Physiotherapy

STUDY DESIGN:
Intervention Model Description: Non-randomised comparative trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimming programme (Experimental): Participants allocated to the swimming programme will be invited to complete three short questionnaires to assess general health, back pain, and swimming ability and experience, see Appendix H, I and J. Both the swimming and physiotherapy groups will complete the three outcome measures, the Oswestry low back pain disability index (ODI), the pain self-efficacy questionnaire (PSEQ), and the EQ-5D-3L, before the intervention, after the last appointment and 6 months later. Data will be collected to report participant characteristics: including age, gender, and length of time with LBP. A follow up participant feedback questionnaire will be distributed to the participants in the swimming arm on completion of the programme and 6 months later.
  Interventions: Other: Swimming programme
- Standard Physiotherapy care (Active Comparator): The participants in the physiotherapy arm will attend the physiotherapy department in the hospital. Treatment delivered by the physiotherapist could include exercise, advice, education, and manual therapy; they will be offered up to 6 sessions. Some appointments will be delivered in a cubicle and others in the physiotherapy gym. The time between appointments varied from person to person.
  Interventions: Other: Standard Physiotherapy care

INTERVENTIONS:
Other: Swimming programme — A session plan will be followed, which included aims, objectives, learning outcomes and suggested core aquatic skills and swimming activities under each section. The session will consist of a session brief, a warmup, core aquatic skills, swimming strokes (front crawl, backstroke, breaststroke, and hybrid strokes), a cool down and a session debrief; following the guidance developed in study three.
  Arms: Swimming programme
Other: Standard Physiotherapy care — Treatment delivered by the physiotherapist could include exercise, advice, education, and manual therapy; they will be offered up to 6 sessions.
  Arms: Standard Physiotherapy care

SUMMARY:
Study four: A small scale RCT will be conducted to pilot the swimming lessons developed in study three, to compare the lessons to standard physiotherapy care and to assess the feasibility of conducting a large RCT in the future. The results from this feasibility study will give the researcher some initial feedback on the swimming lessons and will inform and support the development of an RCT in the future; if the initial findings are positive. This will include whether an RCT can be carried out and evaluating recruitment and retention rates, willingness to be randomised, adverse events, outcomes, acceptability and cost analysis.

DETAILED DESCRIPTION:
Low back pain is very common; globally it is the number one cause of disability. National guidelines recommend exercise for the management of back pain; swimming is frequently advised despite little supporting evidence. Swimming is considered to be low impact and might target conditions associated with back pain such as obesity, inactivity, and depression. Swimming lessons are not funded by the NHS, many adults cannot swim and there are no guidelines regarding what type of swimming program to recommend.

This multi-phase mixed methods research project aims to develop a swimming class to be used as a form of rehabilitation for persistent low back pain. There are many barriers to exercise and this can affect uptake and adherence; Study 1 will be an online survey finding out what stops and what encourages people with back pain to go swimming. Some people already use swimming to manage back pain; in Study 2, individuals who use swimming to manage back pain will be interviewed to explore their experience including discussion about swimming stroke and adaptations. The swimming class will be developed in Study 3 using the data from Study 1 and 2 and by consulting physiotherapists, swimming teachers, and patients, through a series of surveys, known as the Delphi method. Study 4 will be a feasibility study; comparing the swimming class developed in Study 3 over 3 weeks to standard physiotherapy care. Data will be collected on the running of the study, outcomes including function and quality of life, with further follow up at on completion of the trial and 6 months. These studies will be carried out at East Kent Hospitals NHS Trust and the Hotel Burstin swimming pool; people with back pain for more than 3 months would be eligible to take part.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were that participants should have experienced CLBP for more than three months, be at least 18 years old and have a small amount of swimming experience.

Exclusion Criteria:

* Exclusion criteria for the study included the following: unable to read or speak English, allergy to chlorine, severe fear of the water, pregnancy, ear infection, already a competent regular swimmer, visual impairment not correctable with glasses, medical contraindication to aquatic exercise or precaution that cannot be resolved. The following back conditions were excluded; red flag conditions (cauda equina syndrome, cancer or tumour related back pain, spinal infection, spinal cord compression, back pain from visceral source), inflammatory back pain, fractures of the spine during the last 6 months, severe spinal stenosis, nerve root compromise causing neurological deficit or constant pain in the leg, back surgery in the last 6 months, and fitted with a spinal cord stimulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Self efficacy questionnaire | Baseline, 3 weeks and 6 months
  10 questions scored on a Likert scale asking the participant how confident they are to do an activity despite the pain.

SECONDARY OUTCOMES:
Oswestry low back pain disability index | Baseline, 3 weeks and 6 months
  This questionnaire is composed of 10 questions with 6 response statements to assess disability
EQ-5D-3L | Baseline, 3 weeks and 6 months
  Measure of health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Mills, PhD, Study Chair — Canterbury Christ Church University
Locations (1):
- David Stephensen, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan but we are happy to share data with other researchers

REFERENCES:
- [Result] Oakes H, de Vivo M, Mills H, Stephensen D. Recommending swimming to people with low back pain: A scoping review. J Bodyw Mov Ther. 2023 Oct;36:274-281. doi: 10.1016/j.jbmt.2023.05.012. Epub 2023 Aug 25. PMID 37949572